CLINICAL TRIAL: NCT02005562
Title: A Randomized Study Comparing the Incidence of Acute Clinical or Subclinical Rejection With Two Dosing Regimens of CellCept in de Novo Renal Transplant Recipients Receiving Induction, Cyclosporine and Brief Steroid Therapy
Brief Title: OPERA Study: A Study of Two Dosing Regimens of CellCept (Mycophenolate Mofetil) in Kidney Transplant Patients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML19912
Record Dates: First submitted 2013-12-04; First posted 2013-12-09 (Estimated); Results first posted 2015-11-11 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-10

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Mycophenolic Acid; Methylprednisolone; Methylprednisolone Hemisuccinate; Cyclosporine

ARMS (2):
- Mycophenolate Mofetil, Adapted Dose (Experimental): Participants received 3 grams (g) mycophenolate mofetil (MMF) tablets per os (p.o.) in divided doses (every 12 hours [q12h]) adapted to mycophenolic acid (MPA) by area under the curve (AUC) beginning on the day of renal transplant, Day 0, or the day before, Day -1, and continuing through Week 52. In addition, induction by interleukin-2R (IL-2R) was administered at Day 0 per standard of care at the site at the investigator's discretion. At 72 hours post-transplantation, participants received cyclosporine 100-1500 nanograms (ng) per (/) milliliter (mL) from Day 0 to (-) Week 4, 800-1200 ng/mL from Week 4 - Week 12 and 500-800 ng/mL from Week 12 - Week 52. Solumedrol 500 mg intravenously (i.v.) was administered before or after the transplantation, and 0.5 milligrams (mg) per kilogram (kg) p.o. daily from Day 1 - Day 7.
  Interventions: Drug: mycophenolate mofetil; Drug: anti-IL-2R; Drug: methylprednisolone; Drug: cyclosporine
- Mycophenolate Mofetil, Fixed Dose (Active Comparator): Participants received 2 g MMF tablets p.o. in divided doses q12h beginning on the day of renal transplant, Day 0, or the day before, Day -1, and continuing through Week 52. In addition, induction by IL-2R was administered at Day 0 per standard of care at the site at the investigators discretion. At 72 hours post-transplantation, participants received cyclosporine 100-1500 ng/mL from Day 0 - Week 4, 800-1200 ng/mL from Week 4 - Week 12 and 500-800 ng/mL from Week 12 - Week 52. Solumedrol 500 mg i.v. was administered before or after the transplantation, and 0.5 mg/kg p.o. daily from Day 1 - Day 7.
  Interventions: Drug: mycophenolate mofetil; Drug: anti-IL-2R; Drug: methylprednisolone; Drug: cyclosporine

INTERVENTIONS:
Drug: mycophenolate mofetil — 3 g p.o. in divided doses q12h beginning on the day of renal transplant, Day 0, or the day before, Day -1, and continuing to Week 52, adapted to MPA by AUC on Weeks 2, 6, 12, 26, and 52 to obtain AUC0-12 of 50 milligrams (mg) multiplied by (*) height (h)/ liter(L).
  Other Names: CellCept
  Arms: Mycophenolate Mofetil, Adapted Dose
Drug: mycophenolate mofetil — 2 g p.o. in divided doses q12h beginning on the day of renal transplant, Day 0, or the day before, Day -1, and continuing to Week 52.
  Other Names: CellCept
  Arms: Mycophenolate Mofetil, Fixed Dose
Drug: anti-IL-2R — Induction by IL-2R was administered at Day 0 per standard of care at the site at the investigators discretion.
Drug: methylprednisolone — 500 mg intravenous (i.v.) was administered before or after the transplantation, and 0.5 mg/kg p.o. daily from Day 1 to Day 7.
  Other Names: Solumedrol
Drug: cyclosporine — 100-1500 nanograms (ng) per milliliter (mL) from Day 0 to Week 4, 800-1200 ng/mL from Week 4 to Week 12 and 500-800 ng/mL from Week 12 to Week 52

SUMMARY:
This study will compare the incidence of acute clinical or subclinical rejection between immunosuppression with CellCept at a starting dose of 3mg po daily with therapeutic drug monitoring and standard immunosuppression with CellCept and a fixed dose of 2g po daily, in kidney transplant recipients receiving induction by anti-IRL2, cyclosporine therapy, and early discontinuation of steroids. Patients will be randomized to one of the two treatment arms. The anticipated time on study treatment is 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, aged 18-75 years of age;
* in receipt of first donor kidney;
* eligible to receive immunosuppressive treatment comprising IRL2, CellCept, cyclosporine and steroids;
* eligible to receive oral treatment from the first day post-transplantation.

Exclusion Criteria:

* patients receiving a second or subsequent kidney transplant, or multi-organ transplant;
* history of malignancy in the last 5 years (except successfully treated squamous cell or basal cell cancer and cervical cancer in situ);
* patients with active hepatitis B and/or hepatitis C, or HIV infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2006-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (21):
- France (21):
  - Bordeaux
  - Brest
  - Clermont-Ferrand
  - Créteil
  - Dijon
  - La Tronche
  - Le Kremlin-Bicêtre
  - Lille
  - Limoges
  - Montpellier
  - Nantes
  - Nice
  - Paris
  - Poitiers
  - Rennes
  - Salouël
  - Strasbourg
  - Suresnes
  - Toulouse
  - Tours
  - Vandœuvre-lès-Nancy

RESULTS

PARTICIPANT FLOW:
Groups:
- Mycophenolate Mofetil, Adapted Dose: Participants received mycophenolate mofetil (MMF), 3 grams (g), tablets or capsules, orally (PO), every 12 hours (q12h) adapted to mycophenolic acid (MPA) by area under the curve (AUC) on Day -1 or Day 0 through Week 52. Participants also received cyclosporine adapted to a 2 hour postdose (C2) level equal to (=) 1000 to 1500 nanograms per milliliter (ng/mL) from Day 0 to Week 4, C2 = 800 to 1200 ng/mL from Weeks 4 to 12, and C2 = 500 to 800 ng/mL from Weeks 12 to 52. Participants also received methylprednisolone 500 milligrams (mg), intravenously (IV), on Day -1 or Day 0, and 0.5 mg per kilogram (mg/kg), PO, daily (maximum daily dose of 60 mg) from Days 1 through 7 (with steroid withdrawal on Day 7). Participants also received anti-interleukin (IL)-2R, per the investigator's discretion.
- Mycophenolate Mofetil, Fixed Dose: Participants received MMF 2 g, tablets or capsules, PO, q12h on Day -1 or Day 0 through Week 52. Participants also received cyclosporine adapted to C2 = 1000 to 1500 ng/mL from Day 0 to Week 4, C2 = 800 to 1200 ng/mL from Weeks 4 to 12, and C2 = 500 to 800 ng/mL from Weeks 12 to 52 and methylprednisolone 500 mg, IV, on Day -1 or Day 0, and 0.5 mg/kg, PO, daily (maximum daily dose of 60 mg) from Days 1 through 7 (with steroid withdrawal on Day 7). Participants also received anti-IL-2R, per the investigator's discretion.
Period: Overall Study
Arm/Group | Mycophenolate Mofetil, Adapted Dose | Mycophenolate Mofetil, Fixed Dose
Started | 127 | 125
Transplanted | 126 | 121
Completed | 115 | 110
Not Completed | 12 | 15
Not completed — Death | 2 | 2
Not completed — Graft loss | 7 | 6
Not completed — Withdrawal by Subject | 2 | 2
Not completed — No transplant | 1 | 4
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population, all randomized renal transplant recipients who received at least 1 dose of MMF.
Groups:
- Mycophenolate Mofetil, Adapted Dose: Participants received MMF, 3 g, tablets or capsules, PO, q12h adapted to MPA by AUC on Day -1 or Day 0 through Week 52. Participants also received cyclosporine adapted to a C2 level = 1000 to 1500 ng/mL from Day 0 to Week 4, C2 = 800 to 1200 ng/mL from Weeks 4 to 12, and C2 = 500 to 800 ng/mL from Weeks 12 to 52. Participants also received methylprednisolone 500 mg, IV, on Day -1 or Day 0, and 0.5 mg/kg, PO, daily (maximum daily dose of 60 mg) from Days 1 through 7 (with steroid withdrawal on Day 7). Participants also received anti-IL-2R, per the investigator's discretion.
- Total: Total of all reporting groups
Arm/Group | Mycophenolate Mofetil, Adapted Dose | Mycophenolate Mofetil, Fixed Dose | Total
Number analyzed (Participants) | 126 | 121 | 247
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (13.2) | 48.5 (13.0) | 48.5 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 43 | 83
  Male | 86 | 78 | 164

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Biopsy-Proven Acute Rejection (BPAR) Before Week 12 or Acute Subclinical Rejection on Protocol Biopsy at Week 12
Description: BPAR was defined as the presence of clinical signs and kidney biopsy that confirmed the rejection before Week 12. Subclinical acute rejection was defined as an increase of serum creatinine at Week 12 strictly less than 10 percent (%) compared to baseline (BL) values and BPAR of Grade greater than or equal to (≥) 1 according to Banff 1997 classification at Week 12.
Time Frame: Week 12
Population: ITT population; only participants with available protocol biopsy at Week 12 and/or a BPAR before Week 12 were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Mycophenolate Mofetil, Adapted Dose | Mycophenolate Mofetil, Fixed Dose
Number analyzed (Participants) | 91 | 86
percentage of participants | 24.2 | 19.8
Statistical Analysis 1: Comparison: Mycophenolate Mofetil, Adapted Dose vs Mycophenolate Mofetil, Fixed Dose; Test type: Superiority or Other; p = 0.479, Chi-squared

2. Secondary Outcome: Serum Creatinine Values [Micromoles Per Liter (µmol/L)]
Description: The mean serum creatinine values at Weeks 2, 4, 6, 12, 16, 26, 39, and 52.
Time Frame: Weeks 2, 4, 6, 12, 16, 26, 39, and 52
Population: ITT population; number (n) = number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Mycophenolate Mofetil, Adapted Dose | Mycophenolate Mofetil, Fixed Dose
Number analyzed (Participants) | 120 | 114
µmol/L
  Week 2 (n=120,114) | 202.41 (144.80) | 201.31 (130.79)
  Week 4 (n=119,113) | 168.92 (95.66) | 174.86 (77.67)
  Week 6 (n=119,113) | 155.74 (84.01) | 158.96 (59.36)
  Week 12 (n=117,112) | 140.80 (53.18) | 147.70 (50.38)
  Week 16 (n=116,112) | 145.48 (83.00) | 148.48 (71.83)
  Week 26 (n=115,112) | 131.73 (42.20) | 143.73 (46.87)
  Week 40 (n=114,108) | 136.24 (45.84) | 141.89 (47.19)
  Week 52 (n=115,110) | 148.62 (124.30) | 144.72 (47.37)
Statistical Analysis 1: Comparison: Mycophenolate Mofetil, Adapted Dose vs Mycophenolate Mofetil, Fixed Dose; Test type: Superiority or Other; p = 0.6736, ANOVA

3. Secondary Outcome: Creatinine Clearance Values Estimated With the Cockcroft-Gault Equation (Milliliters Per Minute [mL/Min])
Description: The mean creatinine clearance values at Weeks 2, 4, 6, 12, 16, 26, 39, and 52 estimated using the Cockcroft-Gault equation.
Time Frame: Weeks 2, 4, 6, 12, 16, 26, 39, and 52
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Mycophenolate Mofetil, Adapted Dose | Mycophenolate Mofetil, Fixed Dose
Number analyzed (Participants) | 120 | 114
mL/min
  Week 2 (n=120,114) | 46.68 (21.05) | 45.26 (18.93)
  Week 4 (n=119,113) | 51.03 (19.17) | 46.73 (18.11)
  Week 6 (n=119,113) | 53.66 (20.94) | 49.77 (19.05)
  Week 12 (n=117,112) | 56.55 (19.40) | 53.01 (20.14)
  Week 16 (n=116,112) | 56.55 (20.14) | 53.49 (19.72)
  Week 26 (n=115,112) | 60.21 (21.35) | 55.18 (20.52)
  Week 40 (n=114,108) | 59.17 (19.86) | 56.81 (21.81)
  Week 52 (n=115,110) | 58.29 (20.42) | 56.45 (22.02)
Statistical Analysis 1: Comparison: Mycophenolate Mofetil, Adapted Dose vs Mycophenolate Mofetil, Fixed Dose; Test type: Superiority or Other; p = 0.2172, ANOVA

4. Secondary Outcome: Creatinine Clearance Values Estimated With the Modification of Diet in Renal Disease (MDRD) Simplified Equation
Description: The mean creatinine clearance values at Weeks 2, 4, 6, 12, 16, 26, 39, and 52 estimated using the MDRD simplified equation. For males, the MDRD simplified equation was defined as MDRD (mL/min/1.73 square meters [m^2]) =186 multiplied by (*) serum creatinine in mg/L raised to the power of (^) -1.154 * age ^ -0.203. For females, the MDRD simplified equation was defined as MDRD (mL/min/1.73 m^2) = males formula * 0.742.
Time Frame: Weeks 2, 4, 6, 12, 16, 26, 39, and 52
Population: ITT population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Mycophenolate Mofetil, Adapted Dose | Mycophenolate Mofetil, Fixed Dose
Number analyzed (Participants) | 120 | 114
mL/min/1.73 m^2
  Week 2 (n=120,114) | 40.61 (19.00) | 39.60 (18.74)
  Week 4 (n=119,113) | 45.02 (16.58) | 41.31 (16.70)
  Week 6 (n=119,113) | 48.12 (19.32) | 44.69 (16.69)
  Week 12 (n=117,112) | 50.93 (16.27) | 47.68 (16.24)
  Week 16 (n=116,112) | 50.93 (17.05) | 48.52 (17.42)
  Week 26 (n=115,112) | 54.22 (16.76) | 49.46 (18.64)
  Week 40 (n=114,108) | 52.23 (15.94) | 50.01 (18.69)
  Week 52 (n=115,110) | 50.82 (16.33) | 48.88 (18.24)
Statistical Analysis 1: Comparison: Mycophenolate Mofetil, Adapted Dose vs Mycophenolate Mofetil, Fixed Dose; Test type: Superiority or Other; p = 0.4770, ANOVA

5. Secondary Outcome: Time to Occurrence of First BPAR Between Day 0 and Week 52 - Percentage of Participants With an Event
Description: BPAR was defined as the presence of clinical signs and kidney biopsy that confirmed the rejection before Week 12. Subclinical acute rejection at Week 12 was included in the analysis. Subclinical acute rejection was defined as an increase of serum creatinine at Week 12 strictly less than 10% compared to BL values and BPAR of Grade ≥1 according to Banff 1997 classification at Week 12. The occurrence of the first BPAR was defined as the time from randomization to the first recorded BPAR between Day 0 and Week 52. The results of protocol biopsies at Week 12 were taken into account. Participants were censored at the date of last treatment, date of last contact or withdrawal, and date of death.
Time Frame: Day 0, Weeks 2, 4, 6, 12, 16, 26, 39, and 52
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Mycophenolate Mofetil, Adapted Dose | Mycophenolate Mofetil, Fixed Dose
Number analyzed (Participants) | 126 | 121
percentage of participants | 24.6 | 14.9

6. Secondary Outcome: Time to Occurrence of First BPAR Between Day 0 and Week 52
Description: as for outcome 5
Time Frame: Day 0, Weeks 2, 4, 6, 12, 16, 26, 39, and 52
Population: ITT population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Mycophenolate Mofetil, Adapted Dose | Mycophenolate Mofetil, Fixed Dose
Number analyzed (Participants) | 126 | 121
days | NA [NA to NA] — Median time to occurrence of first BPAR was not reached as follow-up time was too short to observe enough events for complete data estimation. | NA [NA to NA] — Median time to occurrence of first BPAR was not reached as follow-up time was too short to observe enough events for complete data estimation.
Statistical Analysis 1: Comparison: Mycophenolate Mofetil, Adapted Dose vs Mycophenolate Mofetil, Fixed Dose; Test type: Superiority or Other; p = 0.0764, Log Rank

7. Secondary Outcome: Percentage of Participants With at Least One BPAR at Week 12 and Week 52
Description: BPAR was defined as the presence of clinical signs and kidney biopsy that confirmed the rejection before Week 12. Participants were censored at the date of last treatment, date of last contact or withdrawal, and date of death.
Time Frame: Weeks 12 and 52
Population: ITT population; only participants with at least one assessed biopsy were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Mycophenolate Mofetil, Adapted Dose | Mycophenolate Mofetil, Fixed Dose
Number analyzed (Participants) | 88 | 80
percentage of participants
  Week 12 | 14.1 | 10.0
  Week 52 | 9.1 | 10.0
Statistical Analysis 1: Comparison: Mycophenolate Mofetil, Adapted Dose vs Mycophenolate Mofetil, Fixed Dose; Week 12; Test type: Superiority or Other; p = 0.418, Fisher Exact
Statistical Analysis 2: Comparison: Mycophenolate Mofetil, Adapted Dose vs Mycophenolate Mofetil, Fixed Dose; Week 52; Test type: Superiority or Other; p = 0.841, Fisher Exact

8. Secondary Outcome: Graft Histology - Percentage of Participants With at Least One Borderline Lesion at Week 12 and Week 52
Description: Participants were censored at the date of last treatment, date of last contact or withdrawal, and date of death.
Time Frame: Weeks 12 and 52
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Mycophenolate Mofetil, Adapted Dose | Mycophenolate Mofetil, Fixed Dose
Number analyzed (Participants) | 126 | 121
percentage of participants
  Week 12 | 7.9 | 12.4
  Week 52 | 6.4 | 5.0
Statistical Analysis 1: Comparison: Mycophenolate Mofetil, Adapted Dose vs Mycophenolate Mofetil, Fixed Dose; Week 12; Test type: Superiority or Other; p = 0.245, Fisher Exact
Statistical Analysis 2: Comparison: Mycophenolate Mofetil, Adapted Dose vs Mycophenolate Mofetil, Fixed Dose; Week 52; Test type: Superiority or Other; p = 0.637, Fisher Exact

9. Secondary Outcome: Graft Histology - Percentage of Participants With at Least One Chronic Graft Nephropathy at Week 12 and Week 52
Description: Participants were censored at the date of last treatment, date of last contact or withdrawal, and date of death.
Time Frame: Weeks 12 and 52
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Mycophenolate Mofetil, Adapted Dose | Mycophenolate Mofetil, Fixed Dose
Number analyzed (Participants) | 126 | 121
percentage of participants
  Week 12 | 20.6 | 17.4
  Week 52 | 32.5 | 34.7
Statistical Analysis 1: Comparison: Mycophenolate Mofetil, Adapted Dose vs Mycophenolate Mofetil, Fixed Dose; Test type: Superiority or Other; p = 0.512, Fisher Exact — Mycophenolate Mofetil, Adapted Dose vs. Mycophenolate Mofetil, Fixed Dose at protocol biopsy at Week 12
Statistical Analysis 2: Comparison: Mycophenolate Mofetil, Adapted Dose vs Mycophenolate Mofetil, Fixed Dose; Test type: Superiority or Other; p = 0.718, Fisher Exact — Mycophenolate Mofetil, Adapted Dose vs. Mycophenolate Mofetil, Fixed Dose at protocol biopsy at Week 52

10. Secondary Outcome: Graft Loss - Percentage of Participants With an Event
Description: Graft loss was defined as physical loss (nephrectomy), functional loss [necessitating maintenance dialysis for greater than (>)8 weeks], retransplant or death. Participants were censored at the date of last treatment, date of last contact or withdrawal, and date of death.
Time Frame: Day 0, Weeks 2, 4, 6, 12, 16, 26, 39, and 52
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Mycophenolate Mofetil, Adapted Dose | Mycophenolate Mofetil, Fixed Dose
Number analyzed (Participants) | 126 | 121
percentage of participants | 5.6 | 5.0

11. Secondary Outcome: Time to Graft Loss
Description: The median time, in days, from randomization to graft loss event. Participants were censored at the date of last treatment, date of last contact or withdrawal, and date of death.
Time Frame: Day 0, Weeks 2, 4, 6, 12, 16, 26, 39, and 52
Population: ITT population
Measure: Median (Full Range); unit: days
Arm/Group | Mycophenolate Mofetil, Adapted Dose | Mycophenolate Mofetil, Fixed Dose
Number analyzed (Participants) | 126 | 121
days | NA (NA) [NA to NA] — Median time to graft loss was not reached as follow-up time was too short to observe enough events for complete data estimation. | NA (NA) [NA to NA] — Median time to graft loss was not reached as follow-up time was too short to observe enough events for complete data estimation.
Statistical Analysis 1: Comparison: Mycophenolate Mofetil, Adapted Dose vs Mycophenolate Mofetil, Fixed Dose; Test type: Superiority or Other; p = 0.860, Log Rank

12. Secondary Outcome: Participant Survival
Description: Participants survival was defined as the percentage of participants living with or without a functioning graft between Weeks 0 and 52. Participants were censored at the date of last treatment, date of last contact or withdrawal, and date of death.
Time Frame: Day 0, Weeks 2, 4, 6, 12, 16, 26, 39, and 52
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Mycophenolate Mofetil, Adapted Dose | Mycophenolate Mofetil, Fixed Dose
Number analyzed (Participants) | 126 | 121
percentage of participants | 98.4 | 98.3

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) were recorded from randomization (Day 0) through the end of study (Week 52).
Description: Safety population: all randomized participants administered at least 1 study treatment dose.
Arm/Group | Mycophenolate Mofetil, Adapted Dose | Mycophenolate Mofetil, Fixed Dose
Serious Adverse Events (participants affected / at risk) | 106/127 | 94/125
Other Adverse Events (participants affected / at risk) | 120/127 | 115/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mycophenolate Mofetil, Adapted Dose (N=127) | Mycophenolate Mofetil, Fixed Dose (N=125)
Cytomegalovirus infection (Infections and infestations) | 18 | 7
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 2
Blood creatinine increased (Investigations) | 15 | 10
Kidney transplant rejection (Renal and urinary disorders) | 49 | 39
Renal failure acute (Renal and urinary disorders) | 14 | 11
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Lymphoproliferative disorder (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 3
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 2
Cardiac failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Nodal arrhythmia (Cardiac disorders) | 0 | 1
Tachyarrhyrhmia (Cardiac disorders) | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 1 | 0
Hyperparathyroidism tertiary (Endocrine disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 4
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Aplasia (General disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Extravasation (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 1 | 0
Hyperthermia (General disorders) | 0 | 1
Inflammation (General disorders) | 0 | 1
Oedema (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 2
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cytolytic hepatitis (Hepatobiliary disorders) | 0 | 1
Bacterial pyelonephritis (Infections and infestations) | 2 | 1
Bronchitis (Infections and infestations) | 0 | 2
Bronchitis acute (Infections and infestations) | 0 | 1
Candida sepsis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 2
Gastroenteritis viral (Infections and infestations) | 1 | 1
Helicobacter gastritis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Incision site abscess (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 2 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 1
Otitis externa (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 | 2
Pyelonephritis (Infections and infestations) | 8 | 7
Pyelonephritis acute (Infections and infestations) | 9 | 5
Renal cyst infection (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 2
Septic shock (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 3
Viral infection (Infections and infestations) | 0 | 2
Blood creatinine abnormal (Investigations) | 0 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Benign colonic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Epstein-Barr virus associated lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 2
Migraine (Nervous system disorders) | 0 | 1
Anxiety disorder (Psychiatric disorders) | 0 | 1
Pelvic haematoma (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Anastomotic haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 | 1
Chronic allograft nephropathy (Injury, poisoning and procedural complications) | 1 | 0
Complication of transplanted kidney (Injury, poisoning and procedural complications) | 1 | 0
Graft dysfunction (Injury, poisoning and procedural complications) | 6 | 6
Graft haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Graft ischaemia (Injury, poisoning and procedural complications) | 1 | 0
Graft thrombosis (Injury, poisoning and procedural complications) | 1 | 1
Nephropathy toxic (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Perirenal haematoma (Injury, poisoning and procedural complications) | 1 | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 1
Post procedural infection (Injury, poisoning and procedural complications) | 1 | 0
Renal haematoma (Injury, poisoning and procedural complications) | 0 | 1
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 | 1
Wound evisceration (Injury, poisoning and procedural complications) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rib fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Postrenal failure (Renal and urinary disorders) | 0 | 1
Pyelocaliectasis (Renal and urinary disorders) | 1 | 1
Pyelonephritis chronic (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 1
Renal haematoma (Renal and urinary disorders) | 1 | 1
Renal impairment (Renal and urinary disorders) | 9 | 9
Renal tubular disorder (Renal and urinary disorders) | 1 | 0
Renal tubular necrosis (Renal and urinary disorders) | 2 | 1
Renal vein thrombosis (Renal and urinary disorders) | 1 | 3
Ureteral necrosis (Renal and urinary disorders) | 0 | 2
Ureteric stenosis (Renal and urinary disorders) | 1 | 3
Urinoma (Renal and urinary disorders) | 1 | 0
Vesicoureteric reflux (Renal and urinary disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cellulitis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Catheter removal (Surgical and medical procedures) | 1 | 0
Transurethral prostatectomy (Surgical and medical procedures) | 1 | 0
Anastomotic stenosis (Vascular disorders) | 1 | 0
Aneurysm (Vascular disorders) | 1 | 0
Aneurysm arteriovenous (Vascular disorders) | 1 | 0
Arterial thrombosis (Vascular disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 1
Arteritis (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 3 | 0
Haemorrhagic cyst (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Iliac artery stenosis (Vascular disorders) | 0 | 1
Lymphocele (Vascular disorders) | 1 | 3
Pelvic venous thrombosis (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 3 | 2
Post procedural haemorrhage (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 2 | 0
Venous thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mycophenolate Mofetil, Adapted Dose (N=127) | Mycophenolate Mofetil, Fixed Dose (N=125)
Anaemia (Blood and lymphatic system disorders) | 71 | 62
Leukopenia (Blood and lymphatic system disorders) | 42 | 23
Diarrheoa (Gastrointestinal disorders) | 18 | 6
Oedema peripheral (General disorders) | 27 | 27
Cytomegalovirus infection (Infections and infestations) | 15 | 14
Urinary tract infection (Infections and infestations) | 28 | 31
Graft dysfunction (Injury, poisoning and procedural complications) | 22 | 10
Blood creatinine increased (Investigations) | 7 | 12
Kidney transplant rejection (Renal and urinary disorders) | 7 | 4
Dysuria (Renal and urinary disorders) | 6 | 7
Hypertension (Vascular disorders) | 18 | 22
Iron deficiency anaemia (Blood and lymphatic system disorders) | 4 | 7
Neutropenia (Blood and lymphatic system disorders) | 10 | 12
Abdominal pain upper (Gastrointestinal disorders) | 8 | 5
Gastrointestinal disorder (Gastrointestinal disorders) | 7 | 0
Gingival hypertrophy (Gastrointestinal disorders) | 10 | 6
Pyrexia (General disorders) | 8 | 7
Proteinuria (Renal and urinary disorders) | 9 | 8
Bronchitis (Infections and infestations) | 4 | 7
Herpes simplex (Infections and infestations) | 7 | 2
Dyslipidaemia (Metabolism and nutrition disorders) | 13 | 17
Diabetes mellitus (Metabolism and nutrition disorders) | 16 | 12
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 9
Overweight (Metabolism and nutrition disorders) | 7 | 5
Underweight (Metabolism and nutrition disorders) | 7 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.